CLINICAL TRIAL: NCT05671887
Title: Double Lung Transplant REgistry Aimed for Lung-limited Malignancies (DREAM) - a Prospective Observational Registry Study for Patients Undergoing Lung Transplantation for Medically Refractory Cancers Confined to the Lungs
Brief Title: DREAM: Double Lung Transplant REgistry Aimed for Lung-limited Malignancies
Acronym: DREAM
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Young Kwang Chae, Associate Professor, Northwestern University
Other Study IDs: STU00217958; NU 22L02 (Other: Northwestern university)
Record Dates: First submitted 2022-12-19; First posted 2023-01-05 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer; Bilateral Cancer; Lung Transplant
Keywords: Cancer; Lung Cancer; Bilateral Cancer; Lung Transplant; Double Lung Transplant; Bronchioloalveolar Carcinoma (BAC); Lepidic; Mucinous
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort A: Primary lung cancers: - Examples include invasive mucinous/non-mucinous non-small cell lung cancers and multifocal carcinomas
  Interventions: Procedure: Double Lung Transplantation
- Cohort B: Metastatic cancers to the lung only: - Examples include germ cell tumors, head & neck tumors, colorectal tumors, renal cell tumors
  Interventions: Procedure: Double Lung Transplantation
- Cohort C: Respiratory failure with a history of cancer in the last 5 years: - Examples include, but not limited to interstitial lung disease (ILD), pulmonary fibrosis (idiopathic or secondary), advanced chronic obstructive pulmonary disease (COPD), bronchiectasis, emphysema, cystic fibrosis (CF), emphysema due to alpha-1 antitrypsin deficiency, and pulmonary arterial hypertension (PAH)
  Interventions: Procedure: Double Lung Transplantation

INTERVENTIONS:
Procedure: Double Lung Transplantation — To evaluate outcomes among patients who undergo lung transplantation for treatment of a select group of medically refractory cancers affecting the lungs alone without extrapulmonary nodal and distant metastasis.
  Other Names: Lung Transplantation

SUMMARY:
This is a prospective observational registration trial for patients who undergo lung transplantation for the treatment of the select groups of medically refractory cancers affecting the lungs alone without extrapulmonary nodal and distant metastasis.

DETAILED DESCRIPTION:
Ever since human lung transplantation was first performed in a patient with advanced lung cancer in 1963 [1], it has emerged as a well-established treatment for patients suffering from a variety of end-stage pulmonary diseases. While lung transplant continues to be performed for refractory lung-limited malignancies that do not have extrapulmonary disease [2-6], given the perceived risks of tumor recurrence following transplantation and potentially reduced survival compared to patients with chronic end-stage lung diseases, transplants for cancer constitutes less than 0.5% of all such procedures (www.srtr.org). The need for lung transplantation is not only confined to patients with primary lung cancers. There are unmet needs for patients who have lung-limited metastasis after successful treatment for primary tumors such as sarcomas or colorectal cancer (CRC). Indeed, successful reports of lung transplantation for lung only metastasis that are refractory to standard of care treatment has been demonstrated [3] and proposed by international experts in highly selected patients [6]. Solid organ transplantation for both primary and metastatic cancers has been demonstrated in liver transplantation [7, 8]. While uncommonly performed, for patients with refractory lung cancer or those with concomitant respiratory failure, lung transplantation may be the only treatment option. The 5-year overall survival of patients in some prior reports who underwent double lung transplantation (DLT) for lung cancer was 39-57%[2, 9], compared to those with non-malignant diseases 50-59%[10, 11]. Indeed, lung transplants have been steadily increasing for cancers, as evident in the International Society of Lung Transplantation (ISHLT) [4-6]. However, the reported cases represent heterogeneity in the surgical technique, patient selection, and post-operative management.

This prospective observational registry aims to better understand the long-term outcomes in patients undergoing double lung transplantation for lung-limited cancers in the clinical programs at Northwestern Medicine and participating centers. We aim to study the impact of a standardized approach to patient selection, tumor staging, surgical technique, and post-operative management on the long-term survival following lung transplantation in patients with lung-limited malignancy. Specifically, this study aims to investigate the clinical outcomes of patients who undergo lung transplantation for treatment of a select group of medically refractory cancers affecting the lungs without extrapulmonary metastases. Patients will undergo transplantation if they have failed standard of care treatments and do not have further curative treatment/trials options. Their clinical courses including overall survival, disease-free survival, and graft failure will be monitored as well as the molecular and genetic biomarkers to investigate the correlation with the prognosis.

ELIGIBILITY:
Inclusion Criteria:

Any patient who is undergoing double lung transplantation as part of the clinical program, consents for this prospective observational trial, and has one of the following conditions will be eligible.

* Common Inclusion Criteria

  * Adults of Age ≦ 80
  * Resistant or refractory to or without available standard of care treatment options or experimental treatment options that are known to increase survival outcome
  * Patients without any extrapulmonary disease
  * Patients with good general health with an ability to withstand physiologic stressors and undergo psychosocial evaluation by the Stanford Integrated Psychosocial Assessment for Transplantation (SIPAT) or other assessment tools
  * Patients to meet all other criteria for lung transplantation including insurance approval and United Network for Organ Sharing (UNOS) registration

Inclusion Criteria for Cohort A

* Histologically confirmed selected lung non-small cell lung cancer including but not limited to:

  o according to the International Association for the Study of Lung Cancer (IASLC)/American Thoracic Society (ATS)/European Respiratory Society (ERS) classification

  - Lepidic dominant pattern
* Adenocarcinoma in situ
* Minimally invasive adenocarcinoma
* Non mucinous lepidic predominant invasive adenocarcinoma

  o based on 2015 World Health Organization (WHO) classification of lung tumors including

  - Invasive mucinous adenocarcinoma
* Mixed invasive mucinous and mucinous adenocarcinoma

  * Colloid adenocarcinoma
  * Enteric adenocarcinoma
  * Minimally invasive adenocarcinoma
* Nonmucinous
* Mucinous

  - Preinvasive lesions
* Atypical adenomatous hyperplasia
* Adenocarcinoma in situ

  * Nonmucinous
  * Mucinous
  * based on the 2004 WHO classification of lung tumors including - Bronchioloalveolar carcinoma
* Nonmucinous
* Mucinous
* Mixed nonmucinous and mucinous or indeterminate
* Without any distant metastasis confirmed by standard staging work-up
* Without brain metastasis confirmed by brain imaging
* Without unidentified primary site of cancer

Inclusion Criteria for Cohort B

* Metastatic cancers to lung alone - including but not limited to germ cell tumors, head & neck tumors, colorectal tumors, renal cell tumors, testicular cancer
* Without any other distant metastasis confirmed by standard staging work-up

Inclusion Criteria for Cohort C

* Respiratory failure with a history of cancer in the last 5 years - including, but not limited to interstitial lung disease (ILD), pulmonary fibrosis (idiopathic or secondary), advanced chronic obstructive pulmonary disease (COPD), bronchiectasis, emphysema, cystic fibrosis (CF), emphysema due to alpha-1 antitrypsin deficiency, and pulmonary arterial hypertension (PAH)
* Without any other distant metastasis confirmed by standard staging work-up

Exclusion Criteria:

* Exclusion criteria

  * Adults unable or unwilling to consent
  * Individuals who are not yet adults (infants, children, teenagers)
  * Pregnant women
  * Prisoners
  * Vulnerable Populations
  * Presence of extrapulmonary disease or mediastinal nodal disease at the time of transplant referral
  * Small Cell Cancers
  * Unidentified primary site of cancer for Cohort A
  * Progression of disease or confirmed distant metastases or mediastinal nodal disease at any point during transplantation work-up
  * Medical ineligibility for lung transplantation after multidisciplinary assessment
  * Not a suitable candidate according to the lung transplantation protocol for treatment of lung confined primary or metastatic tumors
* Body mass index more than 35 kg/m2
* Evidence of co-existing malignancies for Cohort A
* Untreatable significant dysfunction of another major organ system including heart, liver, kidney, or brain unless combined organ transplantation can be performed
* Uncorrected atherosclerotic disease with suspected or confirmed end-organ ischemia or dysfunction and/or coronary artery disease not amenable to revascularization
* Uncorrectable bleeding diathesis
* Evidence of active Mycobacterium tuberculosis infection
* Significant chest wall or spinal deformity expected to cause severe restriction after transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational registration trial for patients who undergo lung transplantation using cadaveric organs for medically refractory cancers affecting the lungs alone and without extrapulmonary metastasis after meeting the inclusion criteria of the clinical program at Northwestern Medicine and participating centers.
  Essential Clinical Criteria:
  1. The tumor should be without any extrapulmonary metastasis as determined by standard of care diagnostic and staging workup.
  2. All standard of care or experimental oncological treatments known to improve survival should have failed or deemed infeasible
  3. Patients should meet the general criteria for lung transplant evaluation and listing
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) rate | 30-day
overall survival (OS) rate | 90-day
disease-free survival (DFS) rate | 30-day
disease-free survival (DFS) rate | 90-day
allograft rejection (AR) rate | 30-day
allograft rejection (AR) rate | 90-day
allograft survival (AS) rate | 30-day
allograft survival (AS) rate | 90-day

SECONDARY OUTCOMES:
overall survival (OS) rate | 6-month, 1-year, 3-year, and 5-year
disease-free survival (DFS) rate | 6-month, 1-year, 3-year, and 5-year
allograft rejection (AR) rate | 6-month, 1-year, 3-year, and 5-year
allograft survival (AS) rate | 6-month, 1-year, 3-year, and 5-year
Major post-transplantation morbidity (MPTM) | 6-month, 1-year, 3-year, and 5-year
  including acute kidney failure requiring continuous renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Young Chae, MD MPH MBA, Principal Investigator — Northwestern University; Ankit Bharat, MD, Principal Investigator — Northwestern University; Rade Tomic, MD, Principal Investigator — Northwestern University
Locations (1):
- Thoracic Surgery, Canning Thoracic Institute (Northwestern Memorial Hospital), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bharat A, Machuca TN, Querrey M, Kurihara C, Garza-Castillon R Jr, Kim S, Manerikar A, Pelaez A, Pipkin M, Shahmohammadi A, Rackauskas M, Kg SR, Balakrishnan KR, Jindal A, Schaheen L, Hashimi S, Buddhdev B, Arjuna A, Rosso L, Palleschi A, Lang C, Jaksch P, Budinger GRS, Nosotti M, Hoetzenecker K. Early outcomes after lung transplantation for severe COVID-19: a series of the first consecutive cases from four countries. Lancet Respir Med. 2021 May;9(5):487-497. doi: 10.1016/S2213-2600(21)00077-1. Epub 2021 Mar 31. PMID 33811829
- [Background] Van Raemdonck D, Vos R, Yserbyt J, Decaluwe H, De Leyn P, Verleden GM. Lung cancer: a rare indication for, but frequent complication after lung transplantation. J Thorac Dis. 2016 Nov;8(Suppl 11):S915-S924. doi: 10.21037/jtd.2016.11.05. PMID 27942415
- [Background] Glanville AR, Wilson BE. Lung transplantation for non-small cell lung cancer and multifocal bronchioalveolar cell carcinoma. Lancet Oncol. 2018 Jul;19(7):e351-e358. doi: 10.1016/S1470-2045(18)30297-3. Epub 2018 Jun 29. PMID 30084382
- [Background] Feldman ER, Eagan RT, Schaid DJ. Metastatic bronchioloalveolar carcinoma and metastatic adenocarcinoma of the lung: comparison of clinical manifestations, chemotherapeutic responses, and prognosis. Mayo Clin Proc. 1992 Jan;67(1):27-32. doi: 10.1016/s0025-6196(12)60273-0. PMID 1310129
- [Background] Grover FL, Piantadosi S. Recurrence and survival following resection of bronchioloalveolar carcinoma of the lung--The Lung Cancer Study Group experience. Ann Surg. 1989 Jun;209(6):779-90. doi: 10.1097/00000658-198906000-00016. PMID 2543339
- [Background] Ahmad U, Wang Z, Bryant AS, Kim AW, Kukreja J, Mason DP, Bermudez CA, Detterbeck FC, Boffa DJ. Outcomes for lung transplantation for lung cancer in the United Network for Organ Sharing Registry. Ann Thorac Surg. 2012 Sep;94(3):935-40; discussion 940-1. doi: 10.1016/j.athoracsur.2012.04.069. Epub 2012 Jul 25. PMID 22835555
- [Background] Garver RI Jr, Zorn GL, Wu X, McGiffin DC, Young KR Jr, Pinkard NB. Recurrence of bronchioloalveolar carcinoma in transplanted lungs. N Engl J Med. 1999 Apr 8;340(14):1071-4. doi: 10.1056/NEJM199904083401403. PMID 10194236
- [Background] Paloyan EB, Swinnen LJ, Montoya A, Lonchyna V, Sullivan HJ, Garrity E. Lung transplantation for advanced bronchioloalveolar carcinoma confined to the lungs. Transplantation. 2000 Jun 15;69(11):2446-8. doi: 10.1097/00007890-200006150-00041. PMID 10868657
- [Background] Zorn GL Jr, McGiffin DC, Young KR Jr, Alexander CB, Weill D, Kirklin JK. Pulmonary transplantation for advanced bronchioloalveolar carcinoma. J Thorac Cardiovasc Surg. 2003 Jan;125(1):45-8. doi: 10.1067/mtc.2003.72. PMID 12538984
- [Background] de Perrot M, Chernenko S, Waddell TK, Shargall Y, Pierre AF, Hutcheon M, Keshavjee S. Role of lung transplantation in the treatment of bronchogenic carcinomas for patients with end-stage pulmonary disease. J Clin Oncol. 2004 Nov 1;22(21):4351-6. doi: 10.1200/JCO.2004.12.188. PMID 15514376
- [Background] Weill D, Benden C, Corris PA, Dark JH, Davis RD, Keshavjee S, Lederer DJ, Mulligan MJ, Patterson GA, Singer LG, Snell GI, Verleden GM, Zamora MR, Glanville AR. A consensus document for the selection of lung transplant candidates: 2014--an update from the Pulmonary Transplantation Council of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2015 Jan;34(1):1-15. doi: 10.1016/j.healun.2014.06.014. Epub 2014 Jun 26. PMID 25085497
- [Background] Dueland S, Grut H, Syversveen T, Hagness M, Line PD. Selection criteria related to long-term survival following liver transplantation for colorectal liver metastasis. Am J Transplant. 2020 Feb;20(2):530-537. doi: 10.1111/ajt.15682. Epub 2019 Nov 28. PMID 31674105
- [Background] Hernandez-Alejandro R, Ruffolo LI, Sasaki K, Tomiyama K, Orloff MS, Pineda-Solis K, Nair A, Errigo J, Dokus MK, Cattral M, McGilvray ID, Ghanekar A, Gallinger S, Selzner N, Claasen MPAW, Burkes R, Hashimoto K, Fujiki M, Quintini C, Estfan BN, Kwon CHD, Menon KVN, Aucejo F, Sapisochin G. Recipient and Donor Outcomes After Living-Donor Liver Transplant for Unresectable Colorectal Liver Metastases. JAMA Surg. 2022 Jun 1;157(6):524-530. doi: 10.1001/jamasurg.2022.0300. PMID 35353121